CLINICAL TRIAL: NCT04668547
Title: Embryoscopic Evacuation for Induced Abortion Using TRUCLEAR Hysteroscopic Morcellator System
Brief Title: Embryoscopic Evacuation for Induced Abortion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Oshri Barell (Other)
Responsible Party: Sponsor-Investigator, Oshri Barell, Head of Gynecology, Assuta Ashdod Hospital
Organization: Assuta Ashdod Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 0206-20-AAA
Record Dates: First submitted 2020-12-09; First posted 2020-12-16 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Induced Abortion and Complications of Termination of Pregnancy
Keywords: Abortion Hysteroscopy Morcellation

STUDY DESIGN:
Intervention Model Description: Feasibility Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional arm (Experimental): Single arm, no comparison
  Interventions: Device: Hysteroscopic Embryolysis

INTERVENTIONS:
Device: Hysteroscopic Embryolysis — Hysteroscopic removal of the products of conception for induced abortion using a hysteroscopic morcellator. If this method of induced abortion fails, a traditional Dilation and Curettage procedure is performed

SUMMARY:
The investigators intend to assess if hysteroscopic evacuation of gestational tissue, is possible as a tool for early induced abortion with a hysteroscopic morcellator rather than with a traditional dilation and curettage procedure. The investigators hypothesize that induced abortion under vision with hysteroscopic guidance may provide benefits over the traditional "blind" procedure

DETAILED DESCRIPTION:
Embryoscopy and fetoscopy had been used increasingly in the treatment of missed abortions in the last two decades. This is done simply by transcervical hysteroscopy during pregnancy. The fact that we can directly view the embryo in the gestational sac allows us to document and describe the fetal morphology and to note different anatomical malformations. Phillips et al described in 2001 the use of embryoscpy prior to evacuation of the uterus in early missed abortions in order to diagnose anatomical malformations and to allow sampling of the fetal tissues for genetic testing. The use of fetal tissue obtained in embryoscopy allows for a more accurate genetic testing and diagnosis and reduces the amount of maternal cells in the specimen.

Hysteroscopic morcellation had been used for intrauterine tissue extraction for over 20 years. Hysteroscopic morcellators have been shown to provide rapid and complete resection of polyps, fibroids, uterine septa and retained products of conception. These instruments use a rotating blade and a suction system that allows for removal for the specimen under direct hysteroscopic visualization. When compared with standard resectoscopic technique, the use of hysteroscopic morcellators probably saves time and allows for more complete removal of the specimen.

A feasibility study conducted in our institute showed that the use of the hysteroscopic morcellator for resection of the fetal tissue in early missed abortions is feasible and safe and might prove beneficial over the standard blind Dilatation and curettage currently used to treat this condition. This technique might allow selective targeting of the fetal tissue thus decreasing the damage caused by trauma to the entire uterine cavity. In a recent systematic review the rate of intrauterine adhesions following D&C for missed abortions ranged between 16 to 21 percent. This technique was assessed prior to our study in only one case published in the literature and was found to be feasible, although the authors state that visibility was poor while resecting the implantation site due to high vascularization.

After demonstrating that hysteroscopic morcellation is possible in cases of early missed abortions, we suggest that the procedure will be possible and safe in cases of early induced abortions, with similar potential benefits.

In this pilot feasibility study, we hypothesize that the Truclear Elite tissue removal system will be able to achieve full evacuation of the uterine cavity. Performed under direct visualization and focused only on the implantation site, thus reducing the potential for further intrauterine adhesions.

This study is a prospective trial. All patients reffered for induced abortion by dilatation and curettage with a gestational age of under 9 weeks in Assuta Ashdod University Hospital that fit the inclusion criteria will be offered to participate.

Two hours prior to the procedure, patients without contraindications can receive cervical preparation with misoprostol 400mcg sublingual.

In theatre under general anesthesia The cervix can be dilated up to an 8 Hegar. Embryoscopy with the TRUCLEAR Elite hysteroscopic morcellation system will be performed and findings will be recorded on a video and in the data collection sheet. The location of the pregnancy, size and specific embryonic findings will be documented.

Following embryoscopy the system will be activated, and the products of conception will be aspirated. If significant bleeding will obscure the hysteroscopic image, vasopressin can be used. 20 units of vasopressin will be diluted in 100ml of saline and injected into the cervix at four and eight o'clock.

The procedure will be performed under abdominal ultrasound guidance to minimize the possibility of perforation. If visibility will be too poor, the procedure will be abandoned and routine suction curettage will be performed using the abdominal ultrasound for guidance All patients will receive prophylactic antibiotics with doxycycline and a follow up appointment with an us examination will be scheduled 2-4 weeks following the procedure and a routine diagnostic hysteroscopy will also be offered 4-6 weeks following the procedure.

Patients will be recruited from the population of patients referred for dilatation and curettage at Assuta Ashdod University Hospital for induced abortion. The researcher will inform the patient about the study. The purpose of the study and possible complications, advantages and alternatives. Patients will not be cajoled into participating in this study. The Investigator will discuss foreseeable risks involved, as well as potential benefits. Patients who have consented to having their information obtained during the study for analysis of the results will have their confidentiality maintained at all times using a study code as an identifier. The patients will be informed by the Investigator that it is their choice to participate and if they do not participate their medical treatment will not be jeopardized. If the patient chooses to participate, they may withdraw from the study at any time without compromising further medical care. A signed and dated Informed Consent must be obtained by the Investigator from the patient prior to enrolment into this study. The original signed and dated information sheet and patient consent will be kept by the Investigator. A signed copy will be provided to the patient.

Since this is a pilot study designed to test the feasibility of the procedure the sample size will include 10 women. This will allow accurate assessment of the procedure and possible issues that might be related to the procedure.

Data collection plan:

1. Pre-procedural: Age, Ethnicity, Weight, Height, Smoking, Medical, Gynecological and Surgical History, Previous hysteroscopies, Previous D&C. Ultrasound scanning findings, LMP.
2. During hysteroscopy: Findings (video recording of procedure), Blood loss, Volume deficit, Length of procedure, Vision, The need to resort to other methods such as D&C, US (ultrasound) findings at the end of the procedure, complications, US during the procedure (recording)
3. Post-procedure: Surgical complications, Hysteroscopy success and post operative course (time to discharge), Findings on follow up examination and US in 2-4 weeks, Findings on follow up diagnostic hysteroscopy in 4-6 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Women between the ages of 21 years - 45 years inclusive.
2. Referred for dilatation and curettage for induced abortion
3. Confirmed intrauterine pregnancy with gestational age of up to 9 weeks
4. At least one previous normal vaginal delivery with a healthy child
5. Patients are able to provide written consent
6. Patients with no underlying medical conditions

Exclusion Criteria:

1. Inability to consent due to cognitive or language barrier
2. Significant uterine bleeding, fever or incomplete abortion
3. Previous cesarean section
4. Sub-chorionic hematoma, Malformed uterus or Submucosal fibroids
5. Any underlying medical condition requiring medical treatment
6. Documented failed hysteroscopy prior to the current referral

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 10 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Completion of the procedure | During the procedure
  Number of patients that were able to complete the procedure under vision without retained products of conception.

SECONDARY OUTCOMES:
Complications | within 30 days from the procedure
  Number of patients with Uterine perforation, Infection, Bleeding re-hospitalization and other complications according to Dindo-Clavien scale

CONTACTS AND LOCATIONS:
Overall Officials: Oshri Barel, MD, Principal Investigator — Assuta Ashdod Medical Center
Locations (1):
- Assuta Ashdod University Hospital, Ashdod, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Philipp T, Kalousek DK. Transcervical embryoscopy in missed abortion. J Assist Reprod Genet. 2001 May;18(5):285-90. doi: 10.1023/a:1016666301481. PMID 11464580
- [Background] Feichtinger M, Wallner E, Hartmann B, Reiner A, Philipp T. Transcervical embryoscopic and cytogenetic findings reveal distinctive differences in primary and secondary recurrent pregnancy loss. Fertil Steril. 2017 Jan;107(1):144-149. doi: 10.1016/j.fertnstert.2016.09.037. Epub 2016 Oct 12. PMID 27743696
- [Background] Campos-Galindo I, Garcia-Herrero S, Martinez-Conejero JA, Ferro J, Simon C, Rubio C. Molecular analysis of products of conception obtained by hysteroembryoscopy from infertile couples. J Assist Reprod Genet. 2015 May;32(5):839-48. doi: 10.1007/s10815-015-0460-z. Epub 2015 Mar 17. PMID 25779005
- [Background] Shazly SA, Laughlin-Tommaso SK, Breitkopf DM, Hopkins MR, Burnett TL, Green IC, Farrell AM, Murad MH, Famuyide AO. Hysteroscopic Morcellation Versus Resection for the Treatment of Uterine Cavitary Lesions: A Systematic Review and Meta-analysis. J Minim Invasive Gynecol. 2016 Sep-Oct;23(6):867-77. doi: 10.1016/j.jmig.2016.04.013. Epub 2016 May 7. PMID 27164165
- [Background] Hooker A, Fraenk D, Brolmann H, Huirne J. Prevalence of intrauterine adhesions after termination of pregnancy: a systematic review. Eur J Contracept Reprod Health Care. 2016 Aug;21(4):329-35. doi: 10.1080/13625187.2016.1199795. PMID 27436757
- [Background] Harpham M, Abbott J. Use of a hysteroscopic morcellator to resect miscarriage in a woman with recurrent Asherman's syndrome. J Minim Invasive Gynecol. 2014 Nov-Dec;21(6):1118-20. doi: 10.1016/j.jmig.2014.05.006. Epub 2014 May 24. PMID 24865632